CLINICAL TRIAL: NCT05782504
Title: Patient-centered Teleprehabilitation for Women With Breast Cancer: a Feasibility Study
Brief Title: Patient-centered Breast Cancer Teleprehabilitation
Acronym: BC-PREHAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other); Ziekenhuis Oost-Limburg (Other); Hasselt University (Other); Kom Op Tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOTK/2022/12550
Record Dates: First submitted 2023-02-08; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Breast Neoplasms; Surgery
Keywords: Prehabilitation; Teleprehabilitation; Breast cancer surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Longitudinal, single-arm, mixed-methods
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): 4 treatment sessions, each lasting 60 minutes, within a 4-week perioperative period, with 2 preoperative (in the last 2 weeks before surgery) and 2 postoperative (in the first 2 weeks after surgery) sessions.
  Interventions: Behavioral: Patient-centered teleprehabilitation

INTERVENTIONS:
Behavioral: Patient-centered teleprehabilitation — Education about the consequences of stress and low physical activity levels with examples of how improving stress tolerance and physical activity can influence QoL and oncological treatment outcomes.
  Exercise therapy based on shared-decision making and using a patient-centered approach. The goal will be to strive for 150-220 min. of moderate physical activity/week, including a home exercise program (at least 1 session/week) of 30-45 min. moderate aerobic exercise, 20 min. of strength training and 10 min. cool down. The latter is guided by Physitrack software.
  Stress management, including questioning personal stress experiences and perceptions, relevant stressors, and stress coping strategies. Next, 3 different relaxation strategies will be explained. Also, cognitive-emotional approaches to stress management and identification of uplifts will be introduced.
  Motivational interviewing will be used during the whole intervention.

SUMMARY:
Surgery, the cornerstone of most cancer treatments, is associated with considerable postoperative complications. Adjusting patients' health behavior before surgery may have beneficial effects on postoperative outcomes.

Women (n=50) who will undergo breast surgery because of stage I-III breast cancer are eligible. All participants will receive multimodal patient-centered teleprehabilitation comprising of motivational interviewing, education, exercise therapy, and stress management.

DETAILED DESCRIPTION:
Feasibility, participation rate, patient satisfaction, intervention safety, and treatment adherence will be monitored as primary outcomes. Fatigue, pain, quality of life (QoL), physical activity levels, perceived injustice, self-efficacy, and healthcare use are secondary outcomes and will be assessed by self-reported questionnaires at baseline, 0-, 2-, and 6 months post-intervention.

Proof of concept for using telecommunication and exercise therapy in prehabilitation prior to breast cancer surgery is available. We expect the proposed intervention to be feasible and effective at reducing fatigue, pain, perceived injustice, and healthcare use, and at improving treatment adherence, QoL, physical activity levels, and self-efficacy.

Effective prehabilitation interventions can reduce the long-term symptoms that arise/persist beyond treatment completion, improving patients' QoL. By using telecommunication technologies, socio-economic barriers can be reduced, making care accessible to all.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Scheduled for primary breast surgery because of stage I-III breast cancer
* Able to speak and read Dutch fluently

Exclusion Criteria:

* Stage IV breast cancer
* A medical contra-indication for physical activity
* Not being able to access a computer or mobile device at home

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Participation rate | one day before the start of the intervention
  This will be calculated as the ratio of the number of patients participating in the study to the number of patients eligible for study participation. Along with that, the participation rate for each of the secondary outcome measures (see further) at each of the time points (baseline and follow-up) will be recorded.
Patient satisfaction with the teleprehabilitation intervention (feeling of contentment with the intervention) | within one week after completion of the intervention
  This will be assessed using a questionnaire ending with an open question ('To what extent is this what you needed? Please explain your answer') and the possibility to suggest alternative treatment content. Patient satisfaction with teleprehabilitation will also be assessed using in-depth interviews with all study participants.
Incidence of treatment-emergent adverse events (safety and tolerability) | within one week after completion of the intervention
  To examine the safety of the intervention, participants will be asked whether they experienced any side effects or unexpected events associated with the intervention after each treatment session.
Adherence to treatment (compliance rate) | within one week after completion of the intervention
  The compliance rate for the teleprehabilitation sessions will be calculated as the ratio of the number of followed treatment sessions versus the number of planned treatment sessions. Next to the supervised sessions, patients will also have sessions without direct supervision that they will have to carry out themselves at home (i.e., exercise sessions, relaxation exercises, and reading the information leaflet). Patients will be asked to record these unsupervised therapy sessions in a personal logbook. The compliance with these home exercise sessions is calculated as the ratio between the number of sessions performed and the number of sessions prescribed.
Feasibility of teleprehabilitation in the clinical setting by means of focus group discussions with stakeholders | through study completion, an average of 1 year
  The feasibility of the patient-centered teleprehabilitation intervention in the clinical setting will be investigated using focus group discussions with all the involved care providers.

SECONDARY OUTCOMES:
Fatigue (feeling of tiredness or lack of energy) | one day before the start of the intervention, one week after completion of the intervention, 30 days after breast surgery, 6 months after breast surgery
  Fatigue is one of the most debilitating symptoms in patients with breast cancer and is the most commonly included cancer-related symptom in core outcome sets for cancer research. For measuring fatigue, the general fatigue subscale of the Multidimensional Fatigue Inventory (MFI-20), a 20-item self-report instrument, will be used. The Dutch MFI-20 is a valid tool to assess cancer-related fatigue in breast cancer patients receiving oncological treatment. This scale has a score from 20 to 100: higher scores indicate a higher level of fatigue.
Pain (uncomfortable sensations in the body) | one day before the start of the intervention, one week after completion of the intervention, 30 days after breast surgery, 6 months after breast surgery
  The Brief Pain Inventory (BPI) is a 14-item questionnaire developed by the World Health Organization Collaborating Centre for Symptom Evaluation in Cancer Care to assess the worst pain, pain severity, and pain interference in cancer patients over the past week reported on a scale of 0 to 10. Pain interference is measured as the average of the 7 interference items, such as walking, mood, and sleep. The BPI is the most common, reliable, and valid outcome measure to assess pain in cancer patients (Cronbach's a and test-retest reliability score > 0.80).
Quality of Life (the degree to which an individual is healthy, comfortable, and able to participate in or enjoy life events) | one day before the start of the intervention, one week after completion of the intervention, 30 days after breast surgery, 6 months after breast surgery
  The European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) is a 30-item cancer-specific questionnaire developed for the assessment of the quality of life in cancer patients. The EORTC QLQ-C30 is the most commonly used patient-reported outcome in breast cancer studies, has been translated and validated in over 100 languages, and shows acceptable psychometric properties. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Subjective level of physical activity | one day before the start of the intervention, one week after completion of the intervention, 30 days after breast surgery, 6 months after breast surgery
  Physical activity of the participants will be assessed with the short form of the International Physical Activity Questionnaire (IPAQ-SF), which subjectively assesses physical activity over the past 7 days. The Dutch version of the IPAQ shows good reliability and validity.
The feeling of perceived injustice | one day before the start of the intervention, one week after completion of the intervention, 30 days after breast surgery, 6 months after breast surgery
  For measuring the feeling of perceived injustice, the Injustice Experience Questionnaire (IEQ) will be used. Participants have to rate the frequency of 12 different statements on a 5-point Likert scale ranging from 0 (not at all) to 4 (all the time), giving a total score that ranges from 0 to 48. The Dutch version of the IEQ is valid and has good (test-retest) reliability (ICC = 0.86-0.87).
Self-efficacy (self-beliefs to cope with a variety of difficult demands in life) | one day before the start of the intervention, one week after completion of the intervention, 30 days after breast surgery, 6 months after breast surgery
  The General Self-Efficacy Scale is a short 10-item scale for assessing optimistic self-beliefs to cope with a variety of difficult demands in life (such as cancer and its treatment), which is widely used, translated, and validated in many languages. This scale has a score from 0 to 90: a higher number on this scale means higher self-efficacy.
Healthcare and medication use during the study period | one day before the start of the intervention, one week after completion of the intervention, 30 days after breast surgery, 6 months after breast surgery
  The healthcare and medication use during the study period, including the use of co-interventions, will be registered with a modified version of the Medical Consumption Questionnaire. This is a generic instrument for measuring the patients' total medical consumption, including additional diagnostics, healthcare visits, hospitalization, physiotherapy, medication, and aids (prescribed by the general practitioner or purchased by the patients themselves).

CONTACTS AND LOCATIONS:
Overall Officials: Jo Nijs, Prof. Dr, Principal Investigator — Vrije Universiteit Brussel
Locations (2):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Jette, Brussels Capital
  - Ziekenhuis Oost-Limburg, Genk

IPD SHARING:
Plan to Share IPD: No